CLINICAL TRIAL: NCT02224508
Title: Evaluation of a Health Plan Initiative to Mitigate Chronic Opioid Therapy Risks
Acronym: CARE
Status: Completed | Type: Observational
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Other Study IDs: PCORI-1306-02198
Record Dates: First submitted 2014-08-15; First posted 2014-08-25 (Estimated); Results first posted 2017-05-05 (Actual); Last update posted 2017-11-13 (Actual); Status verified 2017-10

CONDITIONS: Drug Use Disorders; Drug Abuse; Drug Addiction; Drug Dependence; Drug Habituation; Pain; Depressive Disorder
MeSH Terms: conditions — Substance-Related Disorders; Pain; Depressive Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Opioid Risk Reduction Initiative: Opioid risk reduction initiative for chronic opioid therapy patients implemented in Group Health integrated group practice clinics.
- Usual Care: Usual care for management of chronic opioid therapy patients implemented in Group Health network care settings.

SUMMARY:
Background: Sixty million American adults suffer from moderate to severe chronic pain. Of these, 5 to 8 million currently use opioids long-term. With increased opioid prescribing for chronic pain, an epidemic of prescription opioid addiction and overdose has arisen. This necessitates action to stem opioid-related morbidity and mortality. Group Health (GH), a large nonprofit health plan, developed and implemented opioid risk reduction strategies for doctors and patients in some, but not all, of its clinics. The risk reduction initiative achieved large opioid dose reductions, near universal documentation of care plans, and marked increases in patient monitoring. Rigorous evaluation of patient outcomes resulting from the opioid risk reduction initiative, incorporating patient perspectives, is needed to guide health care improvement efforts to reduce opioid risks regionally and nationally.

Research goal: The investigators will evaluate a major health plan initiative to reduce risks of long-term opioid use for chronic pain. Starting in 2008, some GH clinics reduced prescribing of high opioid doses. In 2010 the same clinics increased care planning and monitoring of chronic opioid therapy (COT) patients. Our research goal is to evaluate effects of this initiative on health and safety outcomes of COT patients. We will test whether the initiative influenced pain outcomes; patient-reported opioid benefits and problems; and opioid-related adverse events.

Design and Outcomes: The investigators will assess effects of GH's opioid risk reduction initiative among COT patients using opioids long-term. The investigators will compare COT patients from clinics that implemented the initiative with COT patients from care settings that did not implement the initiative. The investigators will use survey data to assess patient-reported outcomes including pain severity, depressive symptoms, and patient perceptions of opioid benefits and problems, including validated measures of prescription opioid use disorder. They will interview and compare 800 COT patients using opioids long-term from clinics that implemented the risk reduction initiative and 800 COT patients from care settings that did not.

Impact: This research will provide an urgently needed, rigorous evaluation of a major risk reduction initiative among COT patients. Evaluation results will guide efforts of health plans, clinicians and patients nationwide to ensure safe, effective and compassionate chronic pain care.

DETAILED DESCRIPTION:
Detailed description not provided

ELIGIBILITY:
Inclusion Criteria:

* Enrolled for at least one year prior to sampling for survey
* Received 70+ days supply of opioids in 2 of 4 quarters, including the most recent 90 days
* Received 45+ days supply of opioids in the other 2 quarters

Exclusion Criteria:

* Received cancer diagnoses, other than non-melanoma skin cancer, at least twice in the prior year
* Received any skilled nursing facility care in the prior year
* Received any hospice care or
* Received any opioids from an oncologist

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is prevalent Chronic Opioid Therapy (COT) patients from Group Health clinics. Our initial goals was to interview and compare 800 COT patients using opioids long-term from clinics that implemented the risk reduction initiative and 800 COT patients from care settings that did not. sample size targets were revised to enroll 950 COT patients from the clinics that implemented the risk reduction initiatives and 650 from the clinics that did not implement the risk reduction initiatives.
Sampling Method: Probability Sample
Enrollment: 1588 (Actual)
Dates: Start 2014-09; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael R VonKorff, ScD, Principal Investigator — Group Health Research Institute

IPD SHARING:
Plan to Share IPD: Yes
A complete, cleaned, de-identified copy of the final dataset used in conducting the final analyses will be made available to other qualified researchers within nine months of the end of the final year of funding upon approval by the Group Health Human Subject's Review Committee.
  Given the complexity of the final dataset, our expectation would be that other researchers using the data would require technical assistance from our research team to understand the data and to employ appropriate methods of data analysis. Or, other researchers may prefer to have us analyze the study data to produce analyses according to their specifications. Since use of the dataset by other investigators, or analyses carried out by us for other researchers, would occur after the grant award period has ended, we will expect necessary funding of technical support, data transfers and/or data analyses to be obtained by the research team requesting access to the final dataset.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Opioid Risk Reduction Initiative | Usual Care
Started | 935 (Number of patients surveyed in intervention segment of the health plan (group practice).) | 653 (Number of patients surveyed in the control segment of the health plan (contracted care).)
Completed | 935 | 653
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Opioid Risk Reduction Initiative: Opioid risk reduction initiatives (dose reduction and then risk stratification and monitoring) for chronic opioid therapy patients implemented in Group Health integrated group practice clinics.
- Total: Total of all reporting groups
Arm/Group | Opioid Risk Reduction Initiative | Usual Care | Total
Number analyzed (Participants) | 935 | 653 | 1588
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 507 | 415 | 922
  >=65 years | 428 | 238 | 666
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.6 (12.1) | 61.0 (12.1) | 62.0 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 589 | 420 | 1009
  Male | 346 | 233 | 579
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 804 | 576 | 1380
  African American | 19 | 3 | 22
  Asian/Pacific Islander | 11 | 4 | 15
  Native American | 7 | 3 | 10
  Multiple or other | 83 | 54 | 137
  Missing | 11 | 13 | 24
Education [Count of Participants; unit: Participants]
  High school graduate or less | 243 | 203 | 446
  Some college or technical school | 436 | 296 | 732
  College graduate or post-college graduate | 255 | 152 | 407
  Missing | 1 | 2 | 3
Mental disorder diagnosis past 36 months [Count of Participants; unit: Participants]
  No | 312 | 230 | 542
  Yes | 623 | 423 | 1046
Alcohol use disorder, past 36 months [Count of Participants; unit: Participants]
  No | 885 | 621 | 1506
  Yes | 50 | 32 | 82
Non-opioid drug use disorder diagnosis past 36 months [Count of Participants; unit: Participants]
  No | 846 | 619 | 1465
  Yes | 89 | 34 | 123
Opioid drug use disorder diagnosis, past 36 months [Count of Participants; unit: Participants]
  No | 834 | 577 | 1411
  Yes | 101 | 76 | 177
Tobacco use disorder diagnosis, past 36 months [Count of Participants; unit: Participants]
  No | 711 | 502 | 1213
  Yes | 224 | 151 | 375
Location in Washington State [Count of Participants; unit: Participants]
  Eastern Washington | 242 | 295 | 537
  Western Washington | 693 | 358 | 1051
Marital status [Count of Participants; unit: Participants]
  Not married | 318 | 214 | 532
  Married | 615 | 438 | 1053
  Missing | 2 | 1 | 3
Charlson Comorbidity Score (past 12 months) [Count of Participants; unit: Participants] — The Charlson Comorbidity Score (Romano version) is assessed from electronic health care data for the year prior to the index date. There are 19 sets of conditions, which prior research has shown predict mortality, that are assessed to develop the Charlson Comorbidity Score. Each set of conditions is assigned a weighted score, depending on the estimated risk of subsequent mortality. The Charlson Comorbidity Score also predicts hospitalization risk. The possible total score ranges from 0 to 37, with higher scores indicating greater comorbidity and higher risk of dying.
  Participants
    0 | 426 | 307 | 733
    1 | 75 | 73 | 148
    2 | 144 | 107 | 251
    3-5 | 195 | 127 | 322
    6 or greater | 95 | 39 | 134
Hepatitis C or cirrhosis diagnosis [Count of Participants; unit: Participants]
  No | 851 | 607 | 1458
  Yes | 84 | 46 | 130
Received excess days supply of 20% or greater in any of past 4 quarters [Count of Participants; unit: Participants]
  No | 734 | 493 | 1227
  Yes | 201 | 160 | 361
Average daily opioid dose in morphine equivalents [Count of Participants; unit: Participants]
  No opioid use | 0 | 2 | 2
  Less than 15 milligrams | 232 | 94 | 326
  15 to less than 50 milligrams | 432 | 296 | 728
  50 to less than 120 milligrams | 199 | 150 | 349
  120 milligrams or greater | 72 | 111 | 183
Continuously enrolled in health plan for past 24 months [Count of Participants; unit: Participants]
  No | 48 | 98 | 146
  Yes | 887 | 555 | 1442
Employment status [Count of Participants; unit: Participants]
  Employed full time/part time | 314 | 223 | 537
  Disabled | 182 | 170 | 352
  Retired | 410 | 245 | 655
  Other | 28 | 15 | 43
  Missing | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Proportion With Prescription Opioid Use Disorder (Defined by DSM5 Criteria).
Description: Proportion with Prescription Opioid Use Disorder, which is defined by multiple indicators of opioid abuse and addiction from 9 criteria in the DSM5 manual of the American Psychiatric Association. In this research, it will be assessed using the Psychiatric Research Interview for Substance and Mental Disorders (PRISM5, Columbia University). Estimates were weighted to account for non-response, with weights based on baseline patient characteristics assessed with electronic health care data available for all chronic opioid therapy patients sampled for the survey. The number analyzed differs from the Participant Flow module due to persons with missing item data who were dropped from this analysis. The numbers with missing items were deemed too few to justify item imputation.
Time Frame: 1 year prior to interview
Population: Prevalent chronic opioid therapy (COT) patients defined as having received at least 70 days supply of opioids in the 90 days prior to sample selection, at least 70 days supply of opioids in at least one of the 3 other quarters in the preceding year, and at least 45 days supply of opioids in the other two quarters.
Measure: Number (95% Confidence Interval); unit: proportion of COT patients
Arm/Group | Opioid Risk Reduction Initiative | Usual Care
Number analyzed (Participants) | 934 | 652
proportion of COT patients | 0.215 [0.189 to 0.244] | 0.239 [0.205 to 0.276]

2. Secondary Outcome: Pain Severity (Intensity, Interference With Activities, Enjoyment): PEG Scale
Description: PEG (Pain - Enjoyment - Interference with General Activities) pain scale consisting of the average of 3 0-10 ratings of pain intensity, interference with activities due to pain, and reduced enjoyment of life due to pain. Estimates were weighted to account for non-response, with weights based on baseline patient characteristics assessed with electronic health care data available for all chronic opioid therapy patients sampled for the survey. The PEG score ranges from 0 to 30, with higher scores indicating greater pain severity. The number analyzed differs from the Participant Flow module due to persons with missing item data who were dropped from this analysis. The numbers with missing items were deemed too few to justify item imputation.
Time Frame: 1 week prior to interview
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Opioid Risk Reduction Initiative | Usual Care
Number analyzed (Participants) | 929 | 647
units on a scale | 5.79 [5.65 to 5.93] | 5.82 [5.65 to 5.99]

3. Secondary Outcome: Depressive Symptoms
Description: Patient Health Questionnaire (PHQ-8) depression scale. The PHQ-8 is estimated by summing the 8 scale items. The total score ranges from 0 to 24, with higher scores indicating greater depression severity. Estimates were weighted to account for non-response, with weights based on baseline patient characteristics assessed with electronic health care data available for all chronic opioid therapy patients sampled for the survey. The number analyzed differs from the Participant Flow module due to persons with missing item data who were dropped from this analysis. The numbers with missing items were deemed too few to justify item imputation.
Time Frame: 2 weeks prior to interview
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Opioid Risk Reduction Initiative | Usual Care
Number analyzed (Participants) | 932 | 652
units on a scale | 7.39 [7.04 to 7.74] | 7.91 [7.45 to 8.37]

ADVERSE EVENTS:
Time Frame: The survey was cross-sectional. The prevalent Chronic Opioid Therapy (COT) patients were assessed at the time they were interviewed. The time frame was the year prior to the interview for prescription opioid use disorder, the two weeks prior to the interview for the depressive symptom scale (PHQ-8), and the prior week for the pain severity scale (PEG).
Description: Since study subjects were not tracked over time, we did not assess adverse events occurring over time. The survey assessment did assess prevalent adverse outcomes relevant to chronic opioid therapy (prescription opioid use disorder, depressive symptoms, pain severity).
Arm/Group | Opioid Risk Reduction Initiative | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/935 | 0/653
Serious Adverse Events (participants affected / at risk) | 0/935 | 0/653
Other Adverse Events (participants affected / at risk) | 0/935 | 0/653

LIMITATIONS AND CAVEATS:
This phase of the evaluation reports after-only survey data comparing prevalent chronic opioid therapy patients who had been exposed or not exposed to the health plan opioid risk reduction initiatives for at least one year.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes